CLINICAL TRIAL: NCT07069855
Title: Nutcracker: Can Almond Nut Consumption Improve Nocturnal Glycaemic Control in Women With Gestational Diabetes Mellitus? A Randomised Controlled Trial
Brief Title: Nutcracker: Can Almond Nut Consumption Improve Nocturnal Glycaemic Control in Women With Gestational Diabetes Mellitus?
Acronym: Nutcracker
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 325804
Record Dates: First submitted 2025-05-12; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; pregnancy nutrition; dietary intervention
MeSH Terms: conditions — Diabetes, Gestational | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond group (Experimental): Participants in the almond group will consume 43 g of almonds daily for 28 days, divided into two equal portions: one in the afternoon and one in the evening.
  Interventions: Other: Almond Snack Intervention for Gestational Diabetes
- Control group (Placebo Comparator): Participants in the control group will consume nut-free snacks (e.g., crackers or savoury biscuits) that are energy-matched to the almond snacks.
  Interventions: Other: Control (placebo) group

INTERVENTIONS:
Other: Almond Snack Intervention for Gestational Diabetes — This intervention involves daily consumption of 43 g of whole almonds, split into two portions (afternoon and evening), for 28 days in pregnant women diagnosed with gestational diabetes who habitually consume evening snacks.
  Arms: Almond group
Other: Control (placebo) group — This control involves the daily consumption of a nut-free snack (2 portions) that reflects a 'typical snack' choice among pregnant women with gestational diabetes. It serves as a comparison to assess the specific impact of almond-based evening snacking on overnight glucose regulation.
  Arms: Control group

SUMMARY:
Gestational diabetes, affecting over one in six births globally, is a growing public health concern. Characterised by high blood glucose, it increases the risk of pregnancy complications and raises the mother's long-term risk of type 2 diabetes. Managing high fasting glucose, which reflects elevated overnight levels, is a key challenge. Night-time snacking-more common in women with gestational diabetes-is linked to higher fasting glucose, but the impact of snack quality is unclear. Almonds have been shown to improve glucose control in non-pregnant adults. This study will test whether almonds, as a night-time snack, can improve overnight glucose levels in pregnant women with gestational diabetes. Findings could support a simple, effective dietary strategy to improve outcomes for mothers and babies worldwide.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is a significant and increasingly prevalent public health concern, affecting over one-sixth of births globally. A key challenge in its management is fasting hyperglycaemia, which may result from elevated nocturnal glucose concentrations. Nocturnal hyperglycaemia has been linked to an increased risk of large-for-gestational-age infants in women with GDM. These women are also more likely to snack at night, a behaviour associated with higher fasting glucose concentrations; however, the impact of snack quality on overnight glucose regulation remains unclear.

Almond consumption has been shown to improve glycaemia in individuals with prediabetes or type 2 diabetes, potentially through mechanisms such as carbohydrate displacement and the beneficial effects of their nutrient profile, particularly magnesium and monounsaturated fats. Despite this, research in pregnant populations-especially those with GDM-is limited.

This study will investigate whether consuming almonds as an evening snack for four weeks improves overnight glucose regulation in women with GDM. Participants will be randomised to receive either almonds or a nut-free, energy-matched control snack. Changes in glucose metabolism will be assessed to determine the potential role of almonds in dietary management of GDM.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 16 years
2. Singleton pregnancy
3. 25 to 31+6 weeks' gestation diagnosed with GDM using a standard clinical 75g oral glucose tolerance test (OGTT), as per the guidelines of the National Institute of Health and Care Excellence (NICE), and had their first post-diagnosis consultation (approx. 7-10 days later). The NICE criteria state that the diagnosis of GDM will be made with one or more glucose concentrations during the OGTT of >5.6 mmol/l in the fasting state; >7.8 mmol/l 2 hours after 75g glucose
4. Planned antenatal care at the same centre
5. GDm-Health (a digital app for the management of diabetes in pregnancy) used as part of their management for GDM
6. Willing and able to give informed consent

Exclusion Criteria:

1. Age under 16 years or over 55 years
2. Multiple pregnancy
3. Non-snack consumers
4. Smokers
5. Women who would work night shifts over the study period
6. Women who have already commenced insulin for the treatment of GDM
7. Allergy or intolerance to nuts
8. Pre-existing medical conditions, including Type 1 or Type 2 diabetes, chronic coronary, renal or bowel disease or history of cholestatic liver disease or pancreatitis. Presence of gastrointestinal disorder or use of a drug which is likely to alter gastrointestinal motility or nutrient absorption, previous bariatric surgery
9. Unwilling or unable to give informed consent

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Mean nocturnal blood glucose (22.00-07.00h) | The primary endpoint will be assessed on day 14 and day 28 of the intervention.

SECONDARY OUTCOMES:
Mean daytime glucose 07.00-22.00h | Assessed on day 14 and day 28 of the intervention.
  Recommended glucose control target 3.5-7.8mmol/L, AUC <6.7mmol/L, AUC <7.8mmol/L
Postprandial blood glucose | Assessed on day 14 and day 28 of the intervention.
  Mean postprandial blood glucose for 1, 2 & 4 hours after dinner.
Glucose variability | Assessed on day 14 and 28 of the intervention.
  Glucose SD, glucose CV
Blood glucose indices | Assessed on day 14 and 28 of the intervention.
  High and low blood glucose indices (HBGI & LBGI)
HbA1c | Assessed on day 0 and day 28 of the intervention.
  Biochemical analysis of maternal blood
Liver function | Assessed on day 0 and day 28 of the intervention.
  Biochemical analysis of maternal blood: gamma-glutamyl transferase (GGT), alanine aminotransferase (ALT), aspartate aminotransferase (AST)
Maternal metabolome (blood) | Assessed on day 0 and day 28 of the intervention.
  Lipid measures, including lipoprotein particles (VLDL subdivided into six subclasses, IDL, LDL subdivided into three subclasses, and HDL subdivided into four subclasses), constituents within each lipoprotein particle type (triglycerides, total cholesterol, free cholesterol and cholesterol ester levels and phospholipid concentrations), fatty acids, amino acids, glycolysis related metabolites, ketone bodies and inflammatory markers.
Maternal weight in kg | Assessed on day 0 and day 28 of the intervention.
  Maternal weight and height will be combined to report BMI in kg/m^2
Dietary intake using questionnaire | Assessed on or around day 0 (x2), day 14 (x 2) and day 28 (x2) of the intervention.
  Assessment of dietary intake using Intake24, a validated digital dietary recall system based on the multiple-pass 24-hour recall
Assessment of appetite on a Likert scale | Assessed on day 0, day 14, and day 28 of the intervention.
  Assessment of appetite on a 1-7 Likert scale (i.e., 1 = Not at all hungry, 7 = Extremely hungry)
Physical activity using accelerometer | Assessed on days 0-28 of the intervention.
  The accelerometer will record physical activity, such as average time spent in moderate, low, and sedentary activity
Stool | May be assessed on days 0, 14 and 28 of the intervention.
  (Optional) may be collected and stored for microbiome analysis
Sleep quality using accelerometer | Assessed on days 0-28 of the intervention.
  The accelerometer will measure sleep quality, such as sleep duration
Course of GDM | Assessed on days 0-28 of the intervention.
  If medication is required for glucose control, such as metformin or insulin (dose, time of initiation)
Mode of delivery | Assessed at delivery.
Acceptability of the intervention using questionnaire | Assessed on day 28 of the intervention.
  A dietary intervention acceptability questionnaire will be used to assess enjoyment, sensory aspects, gastrointestinal effects, palatability, and appetite sensations.
Birthweight | Assessed at delivery.
Neonatal head circumference | Assessed at delivery.
Neonatal sex | Assessed at delivery.
Gestational age | Assessed at delivery.
Neonatal complications | Assessed at delivery.
Maternal complications | Assessed at delivery.
Labour onset checklist | Assessed at delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Sara L White, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: Undecided